CLINICAL TRIAL: NCT03767608
Title: Association Between Irisin, Inflammatory Markers and Metabolic Status in Obese Children With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Instituto Tecnologico y de Estudios Superiores de Monterey (Other)
Responsible Party: Principal Investigator, Leticia Elizondo-Montemayor, Dean of the Clinical Nutrition and Obesity Research Center. School of Medicine TEC Salud. Tecnológico de Monterrey, Instituto Tecnologico y de Estudios Superiores de Monterey
Other Study IDs: AIEMPPDM2SM
Record Dates: First submitted 2018-12-04; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus, Type 2; Pediatric Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and plasma were obtained from blood samples and were stored at -80°C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with type 2 diabetes mellitus: Patients diagnosed with T2DM according to the ADA
- Lean healthy controls: Lean healthy controls

SUMMARY:
The objective of this study was to investigate the association of irisin with inflammatory markers as well with metabolic and anthropometric parameters in children and adolescents with type 2 diabetes mellitus compared with healthy controls.

DETAILED DESCRIPTION:
Mexican children and adolescents previously diagnosed with type 2 diabetes mellitus according to the American Diabetes Association (ADA) criteria were recruited and compared to healthy controls.

The participants will undergo:

* vital signs measurement (systolic and diastolic blood pressure, heart rate, respiratory rate)
* anthropometric variables measurement (BMI, weight, waist circumference, hip circumference, body fat %)
* laboratory studies: glucose, triglycerides, HDL-c, C reactive protein, irisin

After statistical analyses the investigators will compare the relationship of irisin and the inflammatory profile and the anthropometric parameters of diabetic patients versus lean controls.

ELIGIBILITY:
Inclusion Criteria:

• Have been previously diagnosed with T2DM according to the American Diabetes Association (ADA) criteria .

Healthy controls were required to have:

* Normal weight according to the Centers for Disease Control and Prevention (CDC) criteria.
* No metabolic abnormalities on blood samples
* No previously diagnosed cardiometabolic diseases
* Not been using antihypertensive, lipid or glucose lowering medications

Exclusion Criteria:

* Disapproval by the children's physician due to any at-risk medical condition known by the parents
* Use of drugs for high blood pressure, hyperglycemia, or dyslipidemia

Ages: 6 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: 40 Mexican children and adolescents aged 7-17 (20 boys and 20 girls) 20 children and adolescents diagnosed with T2DM and 20 healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2017-01-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Correlation of irisin levels and anthropometric parameters in children with type 2 diabetes mellitus (T2DM) | 1 day
  Correlation of irisin levels and anthropometric parameters in children with T2DM
Correlation of irisin levels and anthropometric parameters in healthy control children | 1 day
  Correlation of irisin levels and anthropometric parameters in healthy control children
Correlation of irisin levels and cytokines levels in children with T2DM | 1 day
  Correlation of irisin levels and cytokines levels in children with T2DM
Correlation of irisin levels and C reactive protein levels in healthy control children | 1 day
  Correlation of irisin levels and C reactive protein levels in healthy control children
Comparison between groups | 1 day
  Compare the correlations of irisin woth anthropometric parameters and INFLAMMATORY MARKERSbetween children diagnosed with T2DM and healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Leticia Elizondo-Montemayor, MD, Principal Investigator — Tecnologico de Monterrey, Escuela de Medicina y Ciencias de la Salud
Locations (1):
- Clinical Nutrition and Obesity Research Center. School of Medicine, TEC Salud, Tecnológico de Monterrey, Monterrey, Nuevo León, Mexico